CLINICAL TRIAL: NCT00946608
Title: Comparative, Randomized, Single-Dose, 3-way Crossover Bioavailability Study of Sandoz Inc. and Schering (Claritin) 10 mg Loratadine Tablets In Healthy Adult Male Volunteers Under Fed and Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability Study of Loratadine 10 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA27842
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Allergy
Keywords: Antihistamine
MeSH Terms: conditions — Hypersensitivity | interventions — Loratadine

ARMS (3):
- 1 (Experimental): Loratadine 10 mg Tablets Under Fasting Conditions (Sandoz, Inc.)
  Interventions: Drug: Loratadine 10 mg Tablets Under Fasting Conditions (Sandoz, Inc.)
- 2 (Experimental): Loratadine 10 mg Tablets Under Fed Conditions (Sandoz, Inc.)
  Interventions: Drug: Loratadine 10 mg Tablets Under Fed Conditions (Sandoz, Inc.)
- 3 (Active Comparator): Claritin (Loratadine) 10 mg Tablets Under Fed Conditions (Schering)
  Interventions: Drug: Claritin (Loratadine) 10 mg Tablets Under Fed Conditions (Schering)

INTERVENTIONS:
Drug: Loratadine 10 mg Tablets Under Fasting Conditions (Sandoz, Inc.)
  Arms: 1
Drug: Loratadine 10 mg Tablets Under Fed Conditions (Sandoz, Inc.)
  Arms: 2
Drug: Claritin (Loratadine) 10 mg Tablets Under Fed Conditions (Schering)
  Arms: 3

SUMMARY:
To demonstrate the relative bioavailability study of Loratadine 10 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 54 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — Early Clinical Research